CLINICAL TRIAL: NCT05513287
Title: Retrospective Analytic Study Will be Performed to Investigate if There Was a Change in the Choice of Anethetic Technique for Casrean Section With Continuation of Covid-19 Pandemic
Brief Title: With Continuity of Covid-19 Pandemic, Have Our Anethetic Choices for Caesrean Section Changed ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shereen salah (Other)
Responsible Party: Sponsor-Investigator, Shereen salah, Resident of anethesia, Minia University
Organization: Minia University (Other)
Other Study IDs: Anesthesia with covid
Record Dates: First submitted 2022-07-24; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal anethesia: group number one which recive spinal anethesia in cesarean section in 2020 and 2021
  Interventions: Other: On the period of covid 19
- General anesthesia: Group number 2 which recive general anathesia in cesarean section in 2020 snd 2021
  Interventions: Other: On the period of covid 19

INTERVENTIONS:
Other: On the period of covid 19 — In 2020 and 2021 covid 19 waves in egypt , the effect of this waves in our anathesia in patient wwho undergo cesarean section

SUMMARY:
This retrospective analytic study will be petformed to investigate if there was a change in the choice of anaethetic technique for caesarean sections with continuation of the COVID-19 pandemic .

DETAILED DESCRIPTION:
The number of regional and general anethesia techniques used with detailed number ofspinals epidurals as well as combined spinal epidurals that were provided .

ELIGIBILITY:
Inclusion criteria:

* pregnant women
* suspected or infected with covid-19
* women undergo cesarean section .

Exclusion criteria:

* normal delivery
* abortion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who have seasran section in 18-45 years old
Study Population: Number of regional and general anethesia used in covid waves
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Type of anethesia | 2020,2021
  Number of general and regional anethesia used in pregnant women
Out come of mother | 2 years 2020,2021
  Number of cases whose admitted to icu post operative

SECONDARY OUTCOMES:
Income of mother | 2020,2021
  Numbers of patient whose suspected or infected with covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided